CLINICAL TRIAL: NCT07382635
Title: Clinical Trial Protocol for Evaluating the Efficacy and Safety of Thoracoabdominal Endoscopic Surgery System in Remote Laparoscopic Surgery for Urology, General Surgery, Gynecology and Thoracic Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Cornerstone Robotics (Industry)
Responsible Party: Sponsor
Other Study IDs: F-00300-003
Record Dates: First submitted 2026-01-27; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer; Esophageal Cancer; Hepatectomy; Radical Hysterectomy
Keywords: distal gastric cancer; radical surgery; colorectal cancer; hepatectomy; radical hysterectomy
MeSH Terms: conditions — Colorectal Neoplasms; Esophageal Neoplasms | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Robot-assisted surgery — Surgery with the Cornerstone Surgical Robot.

SUMMARY:
Evaluation of the Efficacy and Safety of the Thoracoabdominal Endoscopic Surgery System Produced by Shenzhen Cornerstone Robotics Technology Co., Ltd. in Remote Laparoscopic Surgeries for Urology, General Surgery, Gynecology and Thoracic Surgery

DETAILED DESCRIPTION:
This trial adopts a prospective, multicenter, single-arm objective value design.For subjects scheduled to undergo thoracoabdominal endoscopic surgery system-assisted laparoscopic surgeries in the departments of urology, general surgery, gynecology and thoracic surgery, the thoracoabdominal endoscopic surgery system developed by Shenzhen Cornerstone Robotics Technology Co., Ltd. will be used to perform remote laparoscopic surgeries in the above four departments, and the efficacy and safety of the investigational medical device in the treatment of remote laparoscopic surgeries in these four departments will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 80 years;
* Patients confirmed by investigators eligible for surgeries in urology (e.g., partial nephrectomy (transperitoneal/retroperitoneal), radical prostatectomy, pyeloplasty, etc.), general surgery (e.g., distal/radical total gastrectomy for gastric cancer, radical resection for colorectal cancer, hepatectomy/splenectomy, etc.), gynecology (e.g., radical hysterectomy plus pelvic lymphadenectomy, etc.) and thoracic surgery (e.g., segmental/lobectomy, radical esophagectomy, etc.).
* Subjects voluntarily participate in the clinical trial, and subjects or their guardians give informed consent and sign the informed consent form.
* Willing to cooperate with and complete trial follow-ups and relevant examinations.

Exclusion Criteria:

* Need for emergency surgery (e.g. gastric cancer, colorectal cancer combined with perforation, bleeding, obstruction, etc.);
* With other malignancies or a previous history of other malignancies.
* Preoperative imaging suggests that the tumour has distant metastases.
* The patient has a history of relevant surgery or previous history of other malignancy and is judged by the investigator to be unsuitable for enrolment.
* Severe bleeding tendencies or coagulopathic disorders.
* With long-term use of anticoagulant and anti-platelet drugs (anti-platelet aggregation drugs discontinued less than 1 week prior to surgery), history of bleeding disorders or hematopoietic or coagulation disorders.
* Significant immunodeficiency due to underlying illness (e.g. HIV/AIDS) and/or medication (e.g. systemic corticosteroids).
* Other conditions which, in the opinion of the investigator, make participation in this trial inappropriate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients confirmed by investigators eligible for surgeries in urology (e.g., partial nephrectomy (transperitoneal/retroperitoneal), radical prostatectomy, pyeloplasty, etc.), general surgery (e.g., distal/radical total gastrectomy for gastric cancer, radical resection for colorectal cancer, hepatectomy/splenectomy, etc.), gynecology (e.g., radical hysterectomy plus pelvic lymphadenectomy, etc.) and thoracic surgery (e.g., segmental/lobectomy, radical esophagectomy, etc.).
Sampling Method: Non-Probability Sample
Enrollment: 98 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Surgical non-referral rate | during the surgery
  Surgical untransferred is defined as not converted from an experimental medical device assisted method to another surgical device control system assisted, laparoscopic surgery or open surgery.

SECONDARY OUTCOMES:
The surgeon's operating time | during the surgery
  Operative time（minutes）
Intraoperative blood loss | during the surgery
  Estimated blood loss（milliliters，ml）
Length of stay | The patient's total number of days from the day of surgery to discharge was recorded 30 days postoperatively.
  The postoperative day when patients complied with the predefined discharge criteria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lai EC, Tang CN. Long-term Survival Analysis of Robotic Versus Conventional Laparoscopic Hepatectomy for Hepatocellular Carcinoma: A Comparative Study. Surg Laparosc Endosc Percutan Tech. 2016 Apr;26(2):162-6. doi: 10.1097/SLE.0000000000000254. PMID 27031650
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/27031650/